CLINICAL TRIAL: NCT03885700
Title: School Intervention Program to Promote Healthy Lifestyle Among Male Adolescent Students in King Faisal Residential City, Jeddah, Western Region, 2014-15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RJ14/014/J
Record Dates: First submitted 2019-02-12; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Physical Activity; Sedentary Behaviors; Dietary Habits; Obesity
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Feeding Behavior; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: Educational program for 2 months
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Educational program for 2 months — The intervention was suggested based on the recommendations for adolescents' healthy diet and physical activity, it was derived from the 2008 Physical Activity Guidelines for Americans and Dietary Guidelines for Americans, 2010 by the U.S. HHS, Physical activity guidelines for children and adolescents by CPS 2012. The Food Guide Pyramid by the USDA, Nutrition &Healthy Eating by Mayo clinic & CDC website. The program was modified according to the age of the child. This plan was typically pursued in a School-based Intervention to Promote Healthy Lifestyles in Sousse, Tunisia, by Harrabi et al. The 1st month covered the healthy diet & the 2nd month covered the physical activity as follow:
  * 1st & 5th week: A 60-minutesession in health education.
  * 2nd & 6th week: Group counselling.
  * 3rd & 7th week: Students were divided into 8 groups & each group was asked to make presentation about a task related to the topic.
  * 4th & 8th week: Discussing the presentation.
  Arms: intervention group

SUMMARY:
Through a cluster randomized control trial, 148 male adolescents' students were randomly assigned into either intervention group who received an educational program for two months (n=79), or control groups (n=69) who didn't attend the program. The principle outcomes were the changes in physical activities, consumption of healthy diet, sedentary life habits and anthropometric measurements. The outcomes of the intervention group were compared with their own baseline readings, as well as with the readings of the control group.

Rationale:

* Saudi adolescents are in need for more exploration of their health problems and related health behaviors and application of intervention preventive services.
* As a National Guard community medicine resident : I have a major interest in the health of adolescent and in fulfilling the aim of the school health programs of application of interventional preventive service that will target this vulnerable risky group.

Aim:

- Promote healthy life style among National Guard adolescents age group by application of interventional preventive program.

Objectives:

I. To measure physical activity patterns , sedentary behaviors and dietary habit among randomly selected adolescent in intervention and control group at National Guard Schools in Jeddah city 2014-2015.

II. To implement an interventional school promotional program among the school children from the addressed age group in 2014-2015.

III. To measure the effect of the interventional school promotional program among the two groups in relation to demographic, socioeconomic and other factors related to health in 2014-2015 .

DETAILED DESCRIPTION:
- Study design: Cluster randomized control trial.

- Study setting: The National Guard health affairs department is a governmental health-providing facility in Saudi Arabia. It is under the Ministry of the National Guard. The National Guard has created residential cities to accommodate military personnel and their families. These cities provide an independent residence with health services, security education, and related services that support optimal living conditions. The National Guard schools provide education from the nursery level up to high school for both males and females, in cooperation with the Ministry of Education. In Jeddah, the National Guard residential city (King Faisal residential city) is located conveniently near the highway (Al-Haramain highway), which is connected to Makkah and Medina and provides quick access to the National Guard medical city (20 minutes away).

The health services in the residential city have two components: the family medicine practice provided by professional teams in Primary Health Care Clinics, and preventive medicine services with implemented programs and activities. One of the major programs in operation in the community and preventive center is the School Health Program, launched in the residential city in 1995. The health affairs division of the National Guard is always on the lookout for further improvement and the expansion of such programs.

The Ministry of National Guard-Health Affairs division aims to improve the school health programs and related activities and encourages all related interventions that have proven effective to the health of the target populations.

Of the seven schools in the residential city, four are elementary, two are intermediate, and one is a high school. The total number of students is 1473.

- Sample size: From the previous study of adolescent lifestyle, the mean weekly moderate activity METs score of male adolescent school students in Jeddah was 1020.4 METs-min/week, (METs-minute ( Metabolic Equivalent of Task (MET) is the ratio of work metabolic rate to a standard resting metabolic rate of 1 (4.184 kJ) kg 5-h- 5 , 1 MET is considered a resting metabolic rate obtained during quiet sitting ).

The least recommended weekly MET by Canadian physical activity guideline's last update was at least 60 minutes of moderate-intensity physical activity every day = 60 X 7days X 4 METs= 1680 METs-min/week.

The use of Pass 13 computer program to calculate the sample size by difference between the two means gives the following results:

Numeric Results for One-Sided Test. Power Clusters Per Clusters Difference Correlation Deviation Alpha Beta 0.90 8 9 579.500 0.02500 1028.50 0.05 0.09

* Summary Statements: A sample size of 8 clusters per group with 9 individuals per cluster achieves 90% power to detect a difference of 579.500 between the group means, when the standard deviation is 1028.500 and the intracluster correlation is 0.02500 using a One-Sided T-test with a significance level of 0.05.
* Taking 10% for the dropout value gives approximately 80 subjects in each group and a total sample size of 160 subjects.
* Sampling technique:

Since the study is cluster-based, eight clusters were considered for each of the intervention and control group. The eight clusters for each group consisted of two classes from the primary schools; one from the 5thgrade and one from the 6th grade, three from the intermediate level (one class from 1st grade, one from the 2nd grade and one from the 3rd grade intermediate school); and three classes from high school (one class from 1st grade, one from the 2nd grade and one from the 3rd grade high school).

Since there were four elementary schools, two schools were selected using random sampling. One school was chosen for the intervention group (Imam Malik's primary school) and one for the control group (Imam Shafiee's primary school). Of the two intermediate schools, one was assigned by random sampling for the intervention (Imam Qaloon's intermediate school), and the second for the control (Abo Obedah's intermediate school). Since there were only one high school, the intervention and control groups were selected by random sampling from the same school (King Saud High School).

The classes were selected by random sampling. Imam Malik's primary school consisted of two classes in the 5th grade and two in the 6thgrade. Two pieces of paper were taken and wrote the names of the two classes on each of the two papers. One paper was drawn at random to select the class that would participate in the intervention group in the study. The same process was repeated for the 6th grade. Imam Shafiee's primary school also consisted of two classes in each grade. Hence, the same process was repeated to select the two classes that would participate in the control group. Imam Qaloon's intermediate school consisted of only one class in each grade, and the same class was assigned to the intervention group. Abo Obediah's intermediate school had four classes in each grade. Four pieces of paper with the class names written on them were made for each grade, and one class was selected by random sampling to participate in the control group. King Saud's high school had four classes in each grade. Four pieces of paper were made for each grade, and two papers were selected from each grade, one for the intervention group and the second for the control group.

Then the research team (which comprised the medical resident and a nurse) went the selected schools, met the principal of the school, and the administration department, to seek their agreement to apply the proposed interventional program. Copies of the list of students in each class were taken from them.

The names of the students for the selected classes were written on pieces of paper, and ten students were selected by random sampling. On the same day, the selected students were given an informed consent form with their names on it and were asked to obtain their parents' consent. The informed consent form consisted of a description of the study population, the study group, the intervention, and the expected harm and benefit from the intervention, it also contained a space for the parents of the selected students to indicate their willingness to allow the child to participate in the study. The students were asked to bring the forms the next day with their parent's signatures.

On the next day, the informed consent forms were collected. Students who were selected by random sampling but did not agree to participate were replaced by students selected by a second random sampling.

* Tools of the study:

  1. Self-administered questionnaire:

     The Arab Teens Lifestyle Study Questionnaire was designed by Hazzaa M Al-Hazzaa whose consent was sought before using it in the study. The Arab Teens Lifestyle Study Questionnaire is a self-reported questionnaire that measures physical activity patterns, sedentary behaviors, and dietary habits, and it was found to be valid by Al-Hazza in his study, "Convergent Validity of the Arab Teens Lifestyle Study (ATLS) Physical Activity Questionnaire" in 2011.

     The questionnaire was designed to collect information on the frequency, duration, and intensity of a variety of light-, moderate- and vigorous-intensity physical activities during a typical (usual) week. These were assigned metabolic equivalent (MET) values based on the compendium of physical activity. By calculating the total METs-minutes per week spent on each of the physical activities, the participants' levels of physical activity were determined.
  2. My plate:

     My Plate is the nutrition guide published by the United States Department of Agriculture, depicting a plate containing five food groups that are part of an ideal diet and a glass. It is a new tool, which has been proven to be appropriate for any age. Through its simplicity, it serves as a guide to help consumers choose nutritionally balanced meals with the right portion size and make healthy choices.
  3. Body composition analyser:

     Tanita BC 418 segmental body composition analyzer was used as it had been shown to be valid in 2009 by Haroun et al. in their study.

     Other tools included a laptop for PowerPoint educational presentations and educational pamphlets.
* Variables collected using the tools:

Dietary habits, physical activity patterns, sedentary behaviours, weight, Body Mass Index (BMI), fat percentage and fat mass.

- Data collection techniques: The team went to the selected school and the students who had received consent were brought by their teachers to the school clinic room; where, the height of each student was measured using a validated measuring scale. The recorded height and age were then entered into the second scale(Tanita BC 418) that measured weight, BMI, fat percentage and fat mass and printed these values on a piece of paper. After the measurements had been completed, each class was handed the self-administered questionnaire, and the questions were explained and filled one at a time by the students under the team's guide.

At the beginning of the study, a total of five schools were visited, and only 148 students agreed to be enrolled in the study.

The interventional school promotional program was conducted for eight consecutive weeks; while the control group did not receive any intervention for the eight weeks in question.

After two months, the second assessment of the healthy behaviours under the study, the weight, BMI, and body composition in the two groups was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent male students in the 5th grade and higher grades at King Faisal residential city schools in Jeddah.

Exclusion Criteria:

-

Ages: 10 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — male
Enrollment: 148 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of the Total Metabolic equivalents (METs) per week. | 2 months
  * The Arab Teens Lifestyle Study Questionnaire was used to measures physical activity level.
  * This Questionnaire was designed to collect information on the:1- frequency 2- duration 3- intensity of a variety of physical activities during a typical week (e.g brisk walking for 20 minutes 3 times per week).
  * These activities were assigned metabolic equivalent (MET)values based on: the compendium of physical activity 2011.
  * Then for each activity the MET equation was applied, METs-min per week for specific activity = duration in min per day × number of days in which the activity were performed per week × METs of that activity (based on the compendium of physical activity 2011).
  * The total METs per week was calculated by combining the METs for all activities performed by each student in his regular week.
measurement of the percentage of students who met the recommended activity level per week. | 2 months
  * For the cut-off value the method used by Al-Hazzaa in his studies was followed, the minimal recommended physical activity per week is equal to 1680 METs.
  * student that had 1680 METs or higher per week were considered to be met the recommended physical activity per week.
  * student that had less than 1680 METs per week was considered to be physical inactive.
  * the percentage of students who met the recommended activity level per week was calculated.
  * the percentage of students who didn't met the recommended activity level per week was calculated.
body weight measurement. | 2 months
  - Tanita BC 418 was used to measure body weight in kg.
height measurement. | 2 months
  - the height was measured in cm using a validated measuring tape.
Body Mass Index measurement. | 2 months
  * the growth chart used by the Saudi Ministry of Health and which was developed by El Mouzan et al was used to plot the Height and weight on the chart to find the corresponding BMI in Kg/M^2 for each student.
  * the BMI categories for adolescents were defined according to the international definition of children's overweight and obesity developed by Cole et al. in 2000.
body fat mass measurement. | 2 months
  -Tanita BC 418 was used to measure body fat mass in Kg for each student.
body fat percentage measurement. | 2 months
  -Tanita BC 418 was used to measure body fat percentage for each student.
measurement of the frequency of consumption of healthy and unhealthy food in regular week. | 2 months.
  * The Arab Teens Lifestyle Study Questionnaire was used to measure dietary habits , as it asses the frequency of consumption of healthy and unhealthy food during regular week.
  * cut-off values :
  * For breakfast, fruit, vegetables, and milk daily consumption was considered as healthy dieting behavior as recommended by healthy food pyramids.
  * For fast food, the measure of three times or more per week was considered as unhealthy dieting behavior.
  * For soft drinks and remaining factors of unhealthy diet, the cut off value of three times per week or more was considered unhealthy dieting behavior.
  * Percentage of each of the healthy and unhealthy food consumption by students in regular week were calculated.
measurement of the time spent daily in different sedentary behaviors. | 2 months
  * The Arab Teens Lifestyle Study Questionnaire was used to measure the time in minutes spent in sedentary behaviors.
  * the allowed daily screen time per day as recommended by Canadian Sedentary Behavior Guidelines was no more than two hours of screen time per day.
  * percentage of student that exceeded the allowed daily screen time were calculated.